CLINICAL TRIAL: NCT01955343
Title: Immune Response in Lung Cancer
Acronym: IRLC
Status: Completed | Type: Observational
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Marius Zemaitis, Assoc. Professor, Lithuanian University of Health Sciences
Other Study IDs: IRLC-1109
Record Dates: First submitted 2013-09-27; First posted 2013-10-07 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Lung Cancer
Keywords: Immune response; Cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood serum and lung biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lung cancer: Newly diagnosed and untreated non small cell lung cancer patients who underwent surgical resection for NSCLC (pathological stage I-III)
- Control: Subjects who will have surgery due to recurrent spontaneous pneumothorax Patients without lung cancer or other malignancies

SUMMARY:
This study is designed to evaluate the importance of the immune cells localization (distribution) between malignant tumor islets and surrounding stroma and to investigate the associations between these immune cells as well as cytokines and clinicopathological and prognostic factors of non-small cell lung cancer (NSCLC) patients.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) score of 0-1
* Patients with histologically documented non-small cell lung cancer
* Control group - patients without non-small cell lung cancer
* Written (signed) Informed Consent to participate in the study

Exclusion Criteria:

* Any other malignancies within 5 years
* Any unstable systemic disease (including active infections, significant cardiovascular disease)
* Prior chemotherapy or radiotherapy
* Autoimmune disease
* Nursing or pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lithuanian residents who are investigated ant treated in Hospital of Lithuanian University of Health Sciences Kaunas Clinics Department of Pulmonology and Immunology and Department of Heart, thoracic and vascular surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2015-07 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
progression-free survival | one year after enrolment to the study

SECONDARY OUTCOMES:
overall survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Marius Zemaitis, Assoc.Prof., Principal Investigator — Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

REFERENCES:
- [Derived] Jackute J, Zemaitis M, Pranys D, Sitkauskiene B, Miliauskas S, Vaitkiene S, Sakalauskas R. Distribution of M1 and M2 macrophages in tumor islets and stroma in relation to prognosis of non-small cell lung cancer. BMC Immunol. 2018 Jan 24;19(1):3. doi: 10.1186/s12865-018-0241-4. PMID 29361917